CLINICAL TRIAL: NCT02311283
Title: Pilot Study: Urea Cycle Disorders Practice Patterns and Outcomes Assessment
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: UCDC5112
Record Dates: First submitted 2014-09-12; First posted 2014-12-08 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2016-09

CONDITIONS: Urea Cycle Disorders
MeSH Terms: conditions — Urea Cycle Disorders, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine if patients participating in "The Longitudinal Study of Urea Cycle Disorders" are different than participants in the Urea Cycles Disorders Consortium (UCDC) Rare Diseases Clinical Research Network (RDCRN) Contact Registry and to determine if patients are a good source of medical information.

DETAILED DESCRIPTION:
Participants enrolled in the RDCRN UCDC Contact Registry will receive an email inviting them to participate in the study. Interested participants will be directed to the informed consent document. After agreeing to participate, participants will be directed to the study web portal. The study web portal will be developed and maintained by the Data Management and Coordinating Center at the University of South Florida (USF).

Participants will complete several questionnaires about their urea cycle disorder including diagnosis and treatment information and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in UCDC RDCRN Contact Registry
* Patient reported diagnosis of one of the eight UCDs or UCD diagnosis highly likely/pending.

Exclusion Criteria:

* Cases of hyperammonemia caused by an organic acidemia, lysinuric protein intolerance, mitochondrial disorders, congenital lactic acidemia, fatty acid oxidation defects and primary liver disease.
* Individuals with rare and unrelated serious comorbidities, e.g., Down syndrome, intraventricular hemorrhage in the newborn period, and extreme low birth weight (<1,500 grams).
* Inability to provide informed consent and complete surveys

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with urea cycle disorders will be recruited via the RDCRN UCDC Contact Registry. The UCDC contact registry consists of over 300 participants with urea cycle disorders.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Test the feasibility of collecting survey data from the UCDC Contact Registry | Up to one year from study activation.
  Patient-reported survey data will be reviewed for accuracy and feasibility as a reliable data source.
Assess patient reported outcomes on urea cycle relevant dimensions (applied cognition & subjective well-being). | Up to one year from study activation.
  The PROMIS website will be used to assess the accuracy and completeness of patient reported outcomes on urea cycle relevant dimensions.
Validate data on treatment setting (team and organization) and management (diet, pharmacologic management, transplantation) | Up to one year from study activation.
  Patient-reported survey data will be linked with research data collected in clinic for the same patients to validate patient-reported data on treatment setting and disease management.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Krischer, PhD, Study Chair — University of South Florida; Jennifer Seminara, MD, Principal Investigator — Children's National Research Institute; Vera Anastasoaie, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- University of South Florida, Tampa, Florida, United States

REFERENCES:
- See also: Rare Diseases Clinical Research Network UCDC webpage — http://www.rarediseasesnetwork.org/ucdc/